CLINICAL TRIAL: NCT05543928
Title: A Multi-Center Study to Evaluate the Efficacy, Safety and Pharmacokinetics of CTAP101 Extended-release Capsules to Treat Secondary Hyperparathyroidism in Pediatric Subjects of Ages 8 to <18 Years With Stage 3 or 4 Chronic Kidney Disease and Vitamin D Insufficiency
Brief Title: Phase 3 Safety and Efficacy Study of CTAP101 Extended-release Capsules in Children With Secondary Hyperparathyroidism
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: FDA changed the post-marketing requirement necessitating a new study design and protocol.
Sponsor: OPKO Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: CTAP101-CL-3007
Record Dates: First submitted 2022-09-13; First posted 2022-09-16 (Actual); Results first posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Chronic Kidney Disease stage3; Chronic Kidney Disease stage4; Vitamin d Deficiency; Secondary Hyperparathyroidism
MeSH Terms: conditions — Vitamin D Deficiency; Hyperparathyroidism, Secondary

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cohort 1 and Cohort 2 Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Cohort 1 and Cohort 2 CTAP101 Capsule (Experimental)
  Interventions: Drug: CTAP101

INTERVENTIONS:
Drug: CTAP101 — CTAP101 Capsules is an extended-release (ER) oral formulation of calcifediol which was approved as Rayaldee® ER Capsules in June 2016 by the United States (US) Food and Drug Administration (FDA) for the treatment of secondary hyperparathyroidism (SHPT) in adult patients with stage 3 or 4 chronic kidney disease (CKD) and vitamin D insufficiency (VDI), defined as serum total 25-hydroxyvitamin D levels less than 30 ng/mL.
  Arms: Cohort 1 and Cohort 2 CTAP101 Capsule
Drug: Placebo — Placebo
  Arms: Cohort 1 and Cohort 2 Placebo

SUMMARY:
This is a phase 3, multi-center, randomized, double-blind, placebo-controlled study in children with stage 3-4 chronic kidney disease (CKD), secondary hyperparathyroidism (SHPT) and vitamin D insufficiency.

ELIGIBILITY:
Inclusion Criteria:

1. Cohort 1: Be 12 to <18 years of age and have a body weight of ≥40 kg; Cohort 2: be 8 to <12 years of age and have a body weight of ≥20 kg.
2. Be diagnosed with stage 3 to 4 CKD at least six months prior to the screening visit, and have an eGFR of ≥15 to <60 mL/min/1.73m2 at screening.
3. Be without any disease state or physical condition that might impair evaluation of safety or which, in the investigator's opinion, would interfere with study participation, including:

   1. Serum albumin ≤ 3.0 g/dL;
   2. Serum transaminase (ALT or SGPT, AST or SGOT) > 2.5 times the upper limit of normal at screening; and,
   3. Urinary albumin excretion of >3000 mcg/mg creatinine.
4. Exhibit during the initial or, if necessary, a screening visit after washout:

   1. Plasma iPTH >100 pg/mL (stage 3 CKD) or >160 pg/mL (stage 4 CKD)
   2. Serum calcium <9.8 mg/dL (corrected for albumin);
   3. Serum total 25-hydroxyvitamin D <30 ng/mL; and,
   4. Serum phosphorus >2.5 to ≤5.5 mg/dL (12 to <18 years) or ≤6.0 mg/dL (ages 8 to <12 years).
5. If taking calcitriol or other 1α-hydroxylated vitamin D analogs, or cinacalcet, be willing to forgo treatment with these agents for the duration of the study and complete an 8-week washout period prior to commencing treatment in the study.
6. If taking >1,000 mg/day of elemental calcium, discontinue or reduce calcium use and/or use non-calcium based therapies for the duration of the study.
7. If receiving ≤1,700 IU/day nutritional vitamin D (ergocalciferol or cholecalciferol) therapy, must agree to remain on a stable dose during the study.
8. If taking >1,700 IU/day of nutritional vitamin D, must discontinue or decrease the dose to ≤1,700 IU/day, maintain that dose for the duration of the study, and complete an 8-week washout period prior to commencing treatment in the study provided that serum total 25-hydroxyvitamin D is ≥30 ng/mL. The washout period is not necessary if serum total 25-hydroxyvitamin D is <30 ng/mL.
9. If taking any bone modifying treatment that could interfere with study endpoints, must discontinue use of such agent(s) for the duration of the study.
10. Willing and able to comply with study instructions and commit to all clinic visits for the duration of the study.
11. Female subjects of childbearing potential must be neither pregnant nor lactating and must have a negative urine pregnancy test at the first screening visit.
12. All female subjects of childbearing potential and male subjects with female partners of childbearing potential must agree to use effective contraception (eg, implants, injectables, combined oral contraceptives, intrauterine device, sexual abstinence, vasectomy or vasectomized partner) for the duration of the study.
13. Each subject or their legal representative must be able to read, understand and sign the informed consent form (ICF).

Exclusion Criteria:

1. History of or planned kidney transplant or parathyroidectomy.
2. History (prior three months) of serum calcium ≥9.8 mg/dL.
3. Use of bisphosphonate therapy (denosumab) within six months prior to enrollment.
4. Known previous or concomitant serious illness or medical condition, such as malignancy, human immunodeficiency virus, significant gastrointestinal or hepatic disease or cardiovascular event or hepatitis, or physical condition that in the opinion of the investigator may worsen and/or interfere with participation in the study.
5. History of neurological/psychiatric disorder, including psychotic disorder, or any reason which, in the opinion of the investigator makes adherence to a treatment or follow up schedule unlikely.
6. Known or suspected hypersensitivity to any of the constituents of either investigational product.
7. Currently participating in, or has participated in, an interventional/investigational study within 30 days prior to study screening.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2023-01-31 (Actual); Primary Completion 2024-06-19 (Actual); Study Completion 2024-06-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Akhtar Ashfaq, MD, Study Director — OPKO Health
Locations (2):
- United States (2):
  - OPKO Study Site, Columbus, Ohio
  - OPKO Study Site, Greenville, South Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort 1 and Cohort 2 Placebo | Cohort 1 and Cohort 2 CTAP101 Capsule
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The study was terminated before randomization
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 and Cohort 2 Placebo | Cohort 1 and Cohort 2 CTAP101 Capsule | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Race (NIH/OMB)
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Numbers of Subjects Who Attained Mean Decrease in Plasma iPTH of 30% From Baseline
Description: The primary efficacy endpoint is the proportion of subjects in the intent-to- treat (ITT) population (age 8 to <18 years) attaining a mean decrease in plasma iPTH of at least 30% from pre-treatment baseline compared to placebo during the EAP.
Time Frame: 26 weeks
Population: The study was terminated before randomization
Arm/Group | Cohort 1 and Cohort 2 Placebo | Cohort 1 and Cohort 2 CTAP101 Capsule
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Safety and Tolerability
Description: Safety and tolerability will be evaluated in the safety population by AEs, PEs, VS, hematology and laboratory evaluations, and ECGs.
Time Frame: 26 weeks
Population: The study was terminated before randomization
Arm/Group | Cohort 1 and Cohort 2 Placebo | Cohort 1 and Cohort 2 CTAP101 Capsule
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Pharmacokinetic
Description: To assess the pharmacokinetic (PK) profile of 25-hydroxyvitamin D3 after repeated doses of CTAP101 Capsules in pediatric subjects
Time Frame: 26 weeks
Population: The study was terminated before randomization
Arm/Group | Cohort 1 and Cohort 2 Placebo | Cohort 1 and Cohort 2 CTAP101 Capsule
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Level of Serum Total 25-hydroxyvitamin D at ≥30 ng/mL Compared to Placebo
Description: To evaluate the efficacy of repeated dosing with CTAP101 Capsules versus placebo in raising serum total 25-hydroxyvitamin D to ≥30 ng/mL
Time Frame: 26 weeks
Population: The study was terminated before randomization
Arm/Group | Cohort 1 and Cohort 2 Placebo | Cohort 1 and Cohort 2 CTAP101 Capsule
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Plasma iPTH Mean Absolute Changes and Serum Total 25-hydroxyvitamin D
Description: To determine the time courses of mean absolute changes from pre-treatment baseline in serum total 25-hydroxyvitamin D and plasma iPTH during administration of repeated doses of CTAP101 Capsules
Time Frame: 26 weeks
Population: The study was terminated before randomization
Arm/Group | Cohort 1 and Cohort 2 Placebo | Cohort 1 and Cohort 2 CTAP101 Capsule
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Pharmacodynamic Effects of Repeated Doses of CTAP101 Capsules
Description: To assess the PD effects of repeated doses of CTAP101 Capsules versus placebo on mean serum calcium (corrected for albumin), serum phosphorus and serum calcium-times-phosphorus (CaxP) product, and the change in mean urine calcium:creatinine ratio
Time Frame: 26 weeks
Population: The study was terminated before randomization
Arm/Group | Cohort 1 and Cohort 2 Placebo | Cohort 1 and Cohort 2 CTAP101 Capsule
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Incidence of Hypercalcemia and Hyperphosphatemia
Description: To evaluate the safety of CTAP101 Capsules versus placebo with regard to the incidence of hypercalcemia and hyperphosphatemia
Time Frame: 26 weeks
Population: The study was terminated before randomization
Arm/Group | Cohort 1 and Cohort 2 Placebo | Cohort 1 and Cohort 2 CTAP101 Capsule
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: The study was terminated before randomization
Arm/Group | Cohort 1 and Cohort 2 Placebo | Cohort 1 and Cohort 2 CTAP101 Capsule
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-11): https://cdn.clinicaltrials.gov/large-docs/28/NCT05543928/Prot_SAP_000.pdf